CLINICAL TRIAL: NCT05016557
Title: The Muscle Protein Synthetic Response Following the Ingestion of a Single Bolus of Algal Protein When Compared to Fungal Protein in Healthy Young Adults
Brief Title: The Muscle Protein Synthetic Response of Algal and Fungal Protein
Acronym: SCAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 200506/B/01
Record Dates: First submitted 2021-08-17; First posted 2021-08-23 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Muscle Metabolism
Keywords: Amino Acids; Protein metabolism; Resistance exercise; Muscle protein synthesis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mycoprotein (Experimental): Bolus ingestion of mycoprotein providing 25g protein
  Interventions: Dietary Supplement: Protein ingestion
- Spirulina (Experimental): Bolus ingestion of spirulina providing 25g protein
  Interventions: Dietary Supplement: Protein ingestion
- Chlorella (Experimental): Bolus ingestion of chlorella providing 25g protein
  Interventions: Dietary Supplement: Protein ingestion

INTERVENTIONS:
Dietary Supplement: Protein ingestion — Bolus ingestion of 25g protein

SUMMARY:
Dietary protein intake is vital for the maintenance of skeletal muscle mass and health. The production of animal-based proteins sources is associated with growing environmental and ethical challenges. As such, sustainable alternatives are needed. Algae are sustainably produced high-protein sources and it is predicted that algae will become one of the most consumed proteins in the next decades. However, the effects of algae on the stimulation of muscle mass growth are unknown. Therefore, we aim to assess the rate of digestion and absorption, and the effects on muscle growth of two types of algae (spirulina and chlorella) when compared to a sustainable non-animal derived fungal reference protein (mycoprotein), a source known to elicit a robust anabolic response.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 and 30
* Recreationally active (<3 times per week structured resistance exercise training)

Exclusion Criteria:

* Any metabolic impairment
* Any cardiovascular impairment
* High blood pressure (>140/90 mmHg)
* A personal history of epilepsy, seizures or schizophrenia
* Smoking
* Chronic (>1 month) use of over the counter pharmaceuticals
* Chronic (>2 months) use of amino acid or protein supplements
* Allergic to Quorn/mycoprotein or algae products

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-12-19 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Muscle Protein Synthesis | 7.5 hours
  The rate of synthesis of new muscle protein (Fractional Synthetic Rate %/h)

SECONDARY OUTCOMES:
Plasma Amino Acid Kinetics | 7.5 hours
  The rate of appearance of amino acid ingested in the drink
Serum Insulin | 7.5 hours
  Basal and postprandial concentrations of serum insulin
Blood Glucose | 7.5 hours
  Basal and postprandial concentrations of blood glucose
mTOR phosphorylation | 7.5 hours
  The amount of mTOR that has been activated in the muscle cell

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin T Wall, PhD, Principal Investigator — Professor of Nutritional Physiology
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No